CLINICAL TRIAL: NCT04533659
Title: Personalized Behavioral Nutrition Intervention in Older Asian Americans With Type 2 Diabetes
Brief Title: Personalized Behavioral Nutrition Intervention in Older AAs With T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Rutgers Asian Resource Center for Minority Aging Research (RCMAR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20200055H
Record Dates: First submitted 2020-08-24; First posted 2020-08-31 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: Personalized behavioral nutrition; Pilot study; Hybrid randomized clinical trial; Older Asian Americans; Metabolomics approach
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This group will receive 4-week diabetes nutrition education with digital self-monitoring for diet and blood glucose.
  Interventions: Behavioral: ADA-based nutrition education with digital self-monitoring
- Intervention group (Experimental): This group will receive 4-week personalized behavioral nutrition intervention with digital self-monitoring for diet and blood glucose and diabetes nutrition education. Participants will discuss the personalized nutrition change goals and recommendations based on metabolic profiling for assessing dietary patterns.
  Interventions: Behavioral: Personalized Behavioral Nutrition (PBN) intervention group

INTERVENTIONS:
Behavioral: ADA-based nutrition education with digital self-monitoring — Diabetes nutrition education developed by the American Diabetes Association with digital self-monitoring for diet and physical activity
  Arms: Control group
Behavioral: Personalized Behavioral Nutrition (PBN) intervention group — Personalized behavioral nutrition intervention consisting of digital self-monitoring for diet and physical activity, personalized nutrition change goal and recommendation, and diabetes nutrition education developed by ADA
  Arms: Intervention group

SUMMARY:
The rapid growth rate and unique challenges as a new immigrant group call for a better understanding of the social and health needs of the older Asian Americans (AAs) population. Overwhelming numbers of AAs, a fast-growing first-generation immigrant group, suffer from type 2 diabetes (T2D) and its consequences of poorly controlled blood glucose. For the older AAs, there are higher prevalence rates, worse diabetes control, and higher rates of complications due to limited English proficiency and health literacy. Despite the evidence concerning the effects of dietary interventions on glycemic control by well-controlled feeding studies in mainstream Americans, a lack of clinical trials of culturally tailored interventions often imposes serious barriers to translate and implement such fruitful and innovative approaches in individuals from ethnic minority communities such as AAs.

The proposed study will use a randomized, controlled design with a sample of 60 AAs aged 65 years or older. Metabolomics methodologies will be incorporated into this research to provide a global picture of metabolites' responses to personalized behavioral nutrition (PBN) intervention. The study results will obtain the necessary information to conduct a meaningful community-based clinical trial to test the effectiveness of PBN in improving dietary patterns and glycemic control in older AAs.

DETAILED DESCRIPTION:
This study is designed with two aims:

1. to determine if PBN intervention improves glycemic control, weight control, and metabolites profiles compared with the control group.
2. to identify significant factors that influence the relative effectiveness of PBN and the relative acceptability of PBN.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as Asian Americans (Chinese, Korean, or South Asian)
2. Age 65 years or older
3. Residing in the Bexar County area
4. Diagnosed with type 2 diabetes; A1C ≥7.5% within 6 months of screening
5. Expressing a willingness to participate in all aspects of the study over its full course
6. Possession of a smartphone

Exclusion Criteria:

1. Unable to give informed consent
2. People under another diet regime that is different from the ADA recommended diet
3. Physical or mental health conditions that could limit active participation in the study (e.g., severe illness, blindness in both eyes, severe immobility, psychiatric diseases)
4. Hematological condition that would affect A1C assay, e.g., hemolytic anemia, sickle cell anemia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Baseline, 4-week, 8-week
  Change in Glycemic control as assessed by HbA1C levels

SECONDARY OUTCOMES:
Metabolites profiles | Baseline, 4-week
  Change in 302 targeted metabolites profiles (e.g. Aconitic acid, Citric acid, Glycolic acid, Homovanillic acid, 2-ET-3-OH-Propionate, 3-OH-Isobutyrate, 3-OH-Isovalerate, 2-3-OH-Propionate, and Uracil)
Lipids profiles | Baseline, 4-week, 8-week
  Change in lipids profiles (LDL, HDL, total cholesterol, triglycerides) as assessed by serum lipids profiling
Weight | Baseline, 4-week, 8-week
  Change in weight as assessed by the Withings electronic scale
Dietary intake | Over the 4-week
  Daily dietary intake as measured by the Fitbit food log
Physical activity | Over the 4-week
  Daily steps taken as measured by the Fitbit wristband
In-home self-monitoring of blood glucose | Over the 4-week
  Daily blood glucose level as measured by wireless glucometer

CONTACTS AND LOCATIONS:
Overall Officials: Jisook Ko, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Ko J, Wang J, Du Y, Jiwani R, Li C. Personalized Behavioral Nutrition Among Older Asian Americans: Study Protocol. Nurs Res. 2021 Jul-Aug 01;70(4):317-322. doi: 10.1097/NNR.0000000000000514. PMID 34160184